CLINICAL TRIAL: NCT03114410
Title: An Evaluation of Re:MIX: a Teen Pregnancy Prevention Program With Young Parents as Peer Educators, EngenderHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: EngenderHealth (Other); University of Texas at Austin (Other); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer Manlove, Senior Program Area Director, Child Trends
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000033-01-01; TP2AH000033-01-01 (Other Grant/Funding Number: HHS Office of Adolescent Health)
Record Dates: First submitted 2017-03-16; First posted 2017-04-14 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Sexual Behavior; Unprotected Sex
MeSH Terms: conditions — Sexual Behavior; Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re:MIX (Experimental): In the experimental arm, the Re:MIX curriculum was implemented. The Re:MIX curriculum is a comprehensive teen pregnancy prevention consisting of ten hour-long sessions, delivered approximately once per week. The Re:MIX curriculum is taught by a professional health educator, partnered with a young parent educator who is a young parent (aged 18-25).
  Interventions: Behavioral: Re:MIX, a multi-layer comprehensive teen pregnancy prevention intervention aimed at reducing pregnancy and STIs among youth ages 13-17
- Comparison (No Intervention): In the comparison arm, teachers were given the option of implementing the Healthy Youth, Healthy You curriculum (focusing on nutrition, mental health, and fitness) or proceed with "business as usual" (no curriculum).

INTERVENTIONS:
Behavioral: Re:MIX, a multi-layer comprehensive teen pregnancy prevention intervention aimed at reducing pregnancy and STIs among youth ages 13-17 — Re:MIX is a comprehensive in-school health curriculum and teen pregnancy prevention program for adolescents covering a broad range of topics related to sexual health and youth development, including healthy relationships, communication, gender, consent, reproductive anatomy, contraception, sexual decision making, clinics, parenthood, and life planning. Re:MIX also aims to connect students and young parent educators with community resources and service linkages. The Re:MIX curriculum teaches mixed-gender groups of students in grades 8 to 10 to delay sex and use protection if they have sex. A co-facilitation team of young parent educators delivered the information with professional health educators using non-traditional approaches, such as game-based tools, technology, and storytelling. Youth received roughly nine hours and 10 minutes of group sessions during the school day over one semester (55 minutes per week for 10 weeks).
  Arms: Re:MIX

SUMMARY:
This study uses a cluster-level randomized controlled design to evaluate the efficacy of Re:MIX in reducing the incidences of early sexual behavior, unprotected sex, oral sex, pregnancy, and STIs. Re:MIX is a comprehensive in-school health curriculum and teen pregnancy prevention program for adolescents covering a broad range of topics related to sexual health and youth development, including healthy relationships, communication, gender, consent, reproductive anatomy, contraception, sexual decision making, clinics, parenthood, and life planning. Re:MIX also aims to connect students and peer educators with community resources and service linkages. The Re:MIX curriculum teaches mixed-gender groups of students in grades 8 to 10 to delay sex and use protection if they have sex. A co-facilitation team of young parent educators delivered the information with professional health educators using non-traditional approaches, such as game-based tools, technology, and storytelling. Youth received roughly nine hours and 10 minutes of group sessions during the school day over one semester (55 minutes per week for 10 weeks). Participants were in 8th, 9th, and 10th graders attending three public charter schools in Travis County, Texas. Comparison classes either received an alternative program that focused on health, nutrition, and fitness, or business as usual. This study was conducted as a Rigorous Evaluation of New or Innovative Approaches to Prevent Teen Pregnancy funded by the U.S. Department of Health and Human Services' Office of Adolescent Health.

ELIGIBILITY:
Inclusion Criteria:

* Students in 8-10th grade classrooms in three public charter schools in Travis County, Texas

Exclusion Criteria:

* None

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 621 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Ever had sexual intercourse | 12 months after baseline
  Single dichotomous item on self-report questionnaire.
Unprotected sexual intercourse in the past 3 months. | 12 months after baseline
  Single dichotomous item on self-report questionnaire.

SECONDARY OUTCOMES:
Intentions | 3 and 12 months after baseline
  Single dichotomous item on self-report questionnaire measuring intentions to have sex in the next year.
Knowledge | 3 and 12 months after baseline
  Outcome was measured using items on a self-report questionnaire related to knowledge about condoms, STI prevention and birth control efficacy
Attitudes | 3 and 12 months after baseline
  Outcome was measured using items on a self-report questionnaire related to attitudes about gender roles, gender and sexual identities, early sex, condom use, early pregnancy and being a teen parent.
Self-efficacy in avoiding unwanted/unprotected sex and communication with partners | 3 and 12 months after baseline
  Outcome was measured using items on a self-report questionnaire related to self-efficacy in obtaining birth control, negotiating condom use avoiding unwanted sexual contact, asking for, and providing consent and assertive communication.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manlove, PhD, Principal Investigator — Child Trends, Senior Program Area Director; Monica Armendariz, Principal Investigator — EngenderHealth: Project Director/Co-Principal Investigator
Locations (1):
- EngenderHealth, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No